CLINICAL TRIAL: NCT04644705
Title: A 3-part Study to Investigate the Safety and Pharmacokinetics of a Novel Niclosamide Solution as a Treatment Option for COVID-19 in Combination With Camostat
Brief Title: Safety and Pharmacokinetics of a Novel Niclosamide Solution in Combination With Camostat
Acronym: NIC-002
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Charité Research Organisation GmbH (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 201767
Record Dates: First submitted 2020-11-02; First posted 2020-11-25 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Niclosamide

STUDY DESIGN:
Intervention Model Description: Part A is a randomized, double-blinded, placebo-controlled, single ascending dose (SAD) study with 3 planned cohorts.
  Part B consists of two randomized, open-label, two-sequence, two-period crossover cohorts comparing the new niclosamide solution with the marketed chewing tablets.
  Part C is a randomized, double-blinded, placebo-controlled multiple dose study investigating the safety and pharmacokinetics of the combination of niclosamide solution and camostat over a treatment period of 7 days.
Who Masked: Participant, Investigator
Masking Description: This three part study has double-blinded (placebo-controlled) and open-label parts.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Part A: verum niclosamide (Active Comparator): The SAD cohorts are planned as follows:
  Cohort A1: 200 mg (fasted conditions) Cohort A2: 600 mg (fasted conditions) Cohort A3: 1600 mg (fasted and fed conditions)
  Interventions: Drug: Niclosamide
- Part A: placebo to niclosamide (Placebo Comparator): The SAD cohorts are planned as follows:
  Cohort A1: placebo to niclosamide 200 mg (fasted conditions) Cohort A2: placebo to niclosamide 600 mg (fasted conditions) Cohort A3: placebo to niclosamide 1600 mg (fasted and fed conditions)
  Interventions: Drug: Placebo
- Part B: verum as solution (niclosamide) (Active Comparator): Two different crossover designs are chosen. Both are randomized, open-label, two-sequence, two periods crossover designs comparing the new niclosamide solution with the marketed chewing tablets. Planned doses are 1600 mg once daily (oral solution), 2000 mg once daily (chewing tablets) and 500 mg three times daily of both dosage forms.
  Interventions: Drug: Niclosamide
- Part B: verum as chewing tablet (niclosamide) (Active Comparator): Two different crossover designs are chosen. Both are randomized, open-label, two-sequence, two periods crossover designs comparing the new niclosamide solution with the marketed chewing tablets. Planned doses are 1600 mg once daily (oral solution), 2000 mg once daily (chewing tablets) and 500 mg three times daily of both dosage forms.
  Interventions: Drug: Niclosamide
- Part C: verum (niclosamide and camostat) (Active Comparator): Subjects will receive the combination of niclosamide solution (planned 500 mg three times daily) + camostat (600 mg three times daily) or placebo over a treatment period of 7 days. The dose of the niclosamide solution depends on the safety and pharmacokinetic results of Part A and B but will not exceed 500 mg three times daily.
  Interventions: Drug: Niclosamide
- Part C: placebo to niclosamide and camostat (Placebo Comparator): Subjects will receive the combination of niclosamide solution (planned 500 mg three times daily) + camostat (600 mg three times daily) or placebo over a treatment period of 7 days. The dose of the niclosamide solution depends on the safety and pharmacokinetic results of Part A and B but will not exceed 500 mg three times daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Niclosamide — Niclosamide will be applied in various dosage steps, galenic preparations and in combination with camostat
  Arms: Part A: verum niclosamide; Part B: verum as chewing tablet (niclosamide); Part B: verum as solution (niclosamide); Part C: verum (niclosamide and camostat)
Drug: Placebo — placebo to the interventional drug
  Arms: Part A: placebo to niclosamide; Part C: placebo to niclosamide and camostat

SUMMARY:
Niclosamide is a well-established substance that is a promising candidate for a repurposing approach to treat COVID-19. Niclosamide is currently marketed as a chewing tablet for the treatment of intestinal worm infections. The marketed formulation is optimized for minimal drug substance absorption. A niclosamide solution has been developed that is expected to release the drug substance more readily and more reproducibly.

Camostat is approved for oral treatment of chronic pancreatitis and reflux oesophagitis in Japan. Camostat has been shown to effectively block viral replication in a SARS-CoV-2 animal model. Since the mechanisms of actions are different, it was hypothesized that a combination of both substances might have an additive or even synergistic effect in the treatment of COVID-19 patients.

This 3-part study is designed to investigate (1) safety and pharmacokinetics of single ascending doses of the new niclosamide solution after fasted and fed conditions, (2) the relative bioavailability of the niclosamide solution compared to the chewing tablet, and (3) safety and pharmacokinetics of the combination of niclosamide solution and camostat after multiple doses in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects in good health as determined by past medical history
* physical examination, vital signs and safety lab at screening
* between 18 to 45 years of age

Exclusion Criteria:

* Significant illness
* pregnant or lactating women

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2021-05-03 (Actual); Study Completion 2021-05-03 (Actual)

PRIMARY OUTCOMES:
Treatment emergent number of Adverse Events | up to 14 days
  Assessment of severity of an AE will be based on CTCAE Version 5.0
Maximum plasma concentration of niclosamide (µg/ml) | from predose until 24 hours after intervention
  Measurement will start at Day 1
Area Under the Plasma Concentration Time Curve from predose until last detectable concentration of niclosamide(AUC0-last) of niclosamide [µg/ml*h] | from predose until 24 hours after intervention
  Measurement will start at Day 1

SECONDARY OUTCOMES:
Food effect on maximum plasma concentration of niclosamide (µg/ml) | from predose until 24 hours after intervention
  Measurement will start at Day 1 after a standard high fat breakfast
Food effect on Area Under the Plasma Concentration Time Curve from predose until last detectable concentration of niclosamide (AUC0-last) [µg/ml*h] | from predose until 24 hours after intervention
  Measurement will start at Day 1 after a standard high fat breakfast
Maximum plasma concentration of niclosamide (µg/ml) at steady state after multiple dosing | from predose until Day 9
Area Under the Plasma Concentration Time Curve between two dosing intervals (AUC tau ss) of niclosamide [µg/ml*h] at steady state after multiple dosing | from predose until Day 9

CONTACTS AND LOCATIONS:
Overall Officials: Maximilian Posch, Dr. med., Principal Investigator — Charité Research Organisation GmbH
Locations (1):
- Charité Research Organisation GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Walther N, Schultz-Heienbrok R, Stass H, Corman VM, Gassen NC, Muller MA, Drosten C, Witzenrath M, Lee H, Posch MG. Clinical safety and pharmacokinetics of a novel oral niclosamide formulation compared with marketed niclosamide chewing tablets in healthy volunteers: A three-part randomized, double-blind, placebo-controlled trial. PLoS One. 2025 Feb 25;20(2):e0303924. doi: 10.1371/journal.pone.0303924. eCollection 2025. PMID 39999124